CLINICAL TRIAL: NCT03759626
Title: Study of the Impact of Two Health Prevention Strategies on Students in the Auvergne-Rhône Alpes Region (I2S-Health Prevention)
Brief Title: I2S-Health Prevention
Acronym: I2S
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-1101SP
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Secondary School Student in General High School Who Does Not Have a Disability That Does Not Allow a Good Understanding of the Study Requirements
Keywords: alcohol; youth; prevention; comparative study; reflexive model; impulsive model; para-social connection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pupils benefiting from the impulsive intervention (Active Comparator): Secondary school pupils from general secondary schools
  Interventions: Behavioral: Impulsive intervention
- pupils benefiting from the reflective intervention (Active Comparator): Second year students from general high schools.
  Interventions: Behavioral: Reflective Intervention

INTERVENTIONS:
Behavioral: Impulsive intervention — As part of the IMAJe project, a 20 min TV series pilot for teenagers was developed by C. Russel of Washington University : "Tom in the making". The results of the study show that the mere diffusion of this pilot mobilizes the individual's impulsive system described in the theoretical model developed by Strack and Deutsch. 2 different versions have been developed. Both have the same basic story in three acts with the same main characters. Only the last acts vary according to the consequences of alcohol consumption. The first version shows a positive representation of alcoholization, the other highlights the negative consequences generated by this behaviour. Our tool will be the so-called "negative" version of the episode where alcohol consumption causes harmful consequences in the young person's life. Following this 20 min episode, a 25 min debate focusing on the characters in the series will be conducted using a questionnaire grid with 8 questions.
  Arms: pupils benefiting from the impulsive intervention
Behavioral: Reflective Intervention — This intervention uses modules of the "KOTTABOS ®" system produced by the National Association for the Prevention of Alcohol and Addiction 59 (ANPAA) and validated by the Interministerial Mission to Combat Drugs and Drug Addiction (MILT). For young people, this educational tool aims to develop an understanding of the mechanisms of blood alcohol levels, the effects and immediate risks associated with alcohol consumption.
  It encourages individual and collective reflection on the effects of alcohol on physical, cognitive and intellectual abilities in order to increase individual skills in making risk-appropriate behavioural choices. This pedagogical tool is based on a participatory and experimental approach. 5 devices of the "KOTTABOS ®" tool were selected and tested with 2 test groups of adolescents of the same school level as the students in the study.
  Arms: pupils benefiting from the reflective intervention

SUMMARY:
Alcohol is the psychoactive substance most experienced by young people. It benefits from positive representations that are reinforced by marketing strategies where advertisers integrate their products into TV series. Our project takes into account the reflexive and impulsive model developed by Strack & Deutsch (2004). We will compare the impulsive intervention to an educational module based on information and reflection that uses the individual's reflexive system with 30 classes in the Loire and Rhône departments. The intervention framework developed uses a modeling system that includes several concepts that work together. These concepts describe the influence of media messages on young people's opinions and behaviours. Given that the objective is to reduce the positive representations of alcohol among young people by means of an educational module based on information and reflection (reflexive model) and a module based on the impulsive system where the para-social connection is involved. The Alcohol Expectancies Scale will be proposed as a judgment criterion and will be administered before and after the intervention.

DETAILED DESCRIPTION:
Alcohol is recognized as responsible for 50,000 premature deaths per year and as the second most preventable cause of death in France. In adolescence, the brain is in a period of maturation. Many synaptic connections are established making the brain more vulnerable to toxic substances. Alcohol is the psychoactive substance most experienced by young people. In 2015, 40% of adolescents and young adults reported drinking alcohol every week. Advertisers are increasingly integrating their products into popular television series. These representations of alcohol in cultural products bypass existing regulations and make it possible to reach a target group that is difficult to reach through traditional advertising: young people. During a previous research project, the Centre Hygée research team, in partnership with American University, carried out a quantitative and qualitative assessment of the images of alcohol in the media viewed by the young public (IMAJe). Within television series, there are many messages inherent to alcohol consumption. Not only is alcohol twice as prevalent in television series as other beverages, but also, alcohol scenes are mainly based on positive results where alcohol refers to celebration and fun. On the other hand, the regularity and stability of the main characters in the series contribute to the viewer's attachment to the series and its characters. This attachment can lead the adolescent to identify with the situations constructed and exposed by developing a "para-social relationship" with the media characters. This connection influences the viewer's appropriation of the messages. This mode of action on opinions and behaviours is to be related to the impulsive model described by Strack & Deutsch (2004).

The main objective of the project is to reduce the positive representations of alcohol among young people by means of an educational module based on information and reflection (reflexive model) and a module based on the impulsive system where the para-social connection is involved.

The intervention framework developed uses a modeling system that includes several concepts that work together. These concepts describe the influence of media messages on young people's opinions and behaviours. This will take into account 1) variables associated with the adolescent's connection to the series and his characters (para-social connection), 2) variables justifying individual differences such as psychological reactance, 3) sociocultural variables. The Alcohol Expectancies Scale will be used before and after the intervention and is proposed as a primary outcome criterion.

Schoolchildren of the Lyon Academy aged between 15 and 19 years old.

There are currently few successful prevention interventions on alcohol representations among young people. The Centre Hygée proposes an original study because it allows the comparison of two logics of prevention intervention but also because the only mobilization of the impulsive system is little used in the prevention sector. The methodology adopted makes it possible to reach validated and effective conclusions for prevention stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* be enrolled in second grade in one of the high schools included
* Have been informed of the study and have not objected to participating
* To be in a general secondary school of general education, of public status
* To be in a high school located in the Auvergne-Rhône Alpes region.

Exclusion Criteria:

* Having a disability that does not allow a good understanding of the study requirements
* Student who opposed participation in the study
* High school without a general education section
* High school included in another research protocol

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 486 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-05-29 (Estimated); Study Completion 2019-06-29 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption level of reprensentation | month 2
  This main criterion will be measured by the "Alcohol Expectancies Scale" translated into French and validated during our previous IMAJe research project. This scale reflects beliefs about the risks and benefits of excessive alcohol consumption (Grube and Agostellino, 1999).
  This 5-point scale with 1 = "very unlikely" and 5 = "very likely" contains 16 items.

SECONDARY OUTCOMES:
The level of intention to consume alcohol | month 2
  The level of their intention to consume alcohol will be assessed through the selection of items related to this theme in the questionnaire used in the HBSC (Health Behaviour in School Aged Children) survey.
  This 7-point scale with 1 = "no chance" and 7 = "certain" has 2 items.
Alcohol consumers level of representation | month 2
  Representations to alcohol consumers will complement the previous measure. They will be evaluated using a scale proposed in the IMAJe questionnaire that has shown excellent psychometric properties.
  This 5-point scale with 1 = "bad" and 5 = "good" contains 6 items.
level of reactance | month 2
  The level of psychological reactance of individuals will be measured using a validated reactance scale, translated from the Hong's Psychological Reactance Scale (HPRS).
  This 5-point scale with 1 = "not at all" and 5 = "completely" contains 7 items.
level of sensation-seeking of individuals | month 2
  The level of their sensation seeking will be measured via Zuckermann's "Sensation Seeking Scale". This scale is used to identify individuals with psychological sensation-seeking traits.
  This 5-point scale with 1 = "strongly disagree" and 5 = "strongly agree" has 6 items.
level of socio-economic status | month 2
  Adolescents' perceptions of social status will be collected with the "Development and Evaluation of a New Indicator".
  This 5-point scale, with 1 = "very comfortable" and 5 = "not at all comfortable" has only 1 item
Consumption of Television Programming | month 2
  the relationship to media content will be measured using the parasocial connection of individuals via the French version of the parasocial connection scale established by Russel et al.
  This 5-point scale with 1 = "strongly disagree" and 5 = "strongly agree" has 16 items.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Régnier-Denois, Study Director — Institut de Cancérologie Lucien Neuwirth
Locations (3):
- Americain University of Washington, Washington, Massachusetts, United States
- France (2):
  - Mutualité Française de la Loire, Saint-Etienne
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No